CLINICAL TRIAL: NCT03662672
Title: Randomized Controlled Trial of Rib Raising as Early Treatment for Post-operative Ileus
Brief Title: Rib Raising for Post-operative Ileus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Nina Elizabeth Glass, MD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2018001548
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Intestinal Pseudo-Obstruction; Manipulation, Osteopathic; Postoperative Care; Postoperative Nausea and Vomiting; Postoperative Complications; Osteopathic Medicine
MeSH Terms: conditions — Intestinal Pseudo-Obstruction; Postoperative Nausea and Vomiting; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rib-raising Intervention (Experimental): We will do daily rib raising and lumbar release from the 5th thoracic vertebra to the 2nd lumbar vertebra for 2 minutes per side for rib raising and 2 minutes for lumbar release.
  Interventions: Procedure: Rib raising and lumbar release
- Sham Intervention (Sham Comparator): We will do daily sham intervention from the 5th thoracic vertebra to the 2nd lumbar vertebra where we place our hands under the ribs for 2 minutes per side and under the lumbar area for 2 minutes without applying any pressure (or applying pressure into the bed).
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Rib raising and lumbar release — Rib raising per protocol described in arm description.
  Arms: Rib-raising Intervention
Procedure: Sham procedure — Sham procedure per protocol described in arm description
  Arms: Sham Intervention

SUMMARY:
We are conducting a randomized controlled trial the use of rib raising for post-operative ileus. Rib raising is an osteopathic manipulative technique (OMT). We will recruit all patients undergoing major abdominal surgery and once they have been enrolled, we will randomize them to receive daily rib raising or a control technique where we place hands on the back but do not apply any pressure. In preliminary studies, Rib raising has been shown to reduce post-operative ileus and hospital length of stay by up to 50%.

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery (laparotomy, laparoscopy excluding simple laparoscopic appendectomy or laparoscopic cholecystectomy)

Exclusion Criteria:

* Open abdomen for >72 hours
* Prior history of major post-operative complications
* Intolerance to anesthesia
* Co-morbidities including osteoporosis and osteopenia
* Spine or rib fractures
* Pregnancy
* Prisoners
* History of osteopathic manipulation
* Recruitment delayed beyond 48 hours
* Surgeon requested exclusion

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Length of Stay | 0-14 days

SECONDARY OUTCOMES:
Time to first meal | 0-14 days
Time to first flatus | 0-14 days
Time to first bowel movement | 0-14 days
Need for nasogastric tube postop | 0-14 days
Nausea/vomiting postop | 0-14 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baltazar GA, Betler MP, Akella K, Khatri R, Asaro R, Chendrasekhar A. Effect of osteopathic manipulative treatment on incidence of postoperative ileus and hospital length of stay in general surgical patients. J Am Osteopath Assoc. 2013 Mar;113(3):204-9. PMID 23485980
- [Background] Crow WT, Gorodinsky L. Does osteopathic manipulative treatment (OMT) improves outcomes in patients who develop postoperative ileus: A retrospective chart review. International Journal of Osteopathic Medicine. 2009;12(1):32-7.
- [Background] Herrmann EP. Postoperative adynamic ileus: its prevention and treatment by osteopathic manipulation. The DO. 1965;6(2):163-4.